CLINICAL TRIAL: NCT00584493
Title: Treatment Use Study of CP-675,206 for Advanced Melanoma
Brief Title: Treatment Use Study for Advanced Melanoma.
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Other Study IDs: A3671028
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-12

CONDITIONS: Advanced Unresectable Melanoma
MeSH Terms: interventions — tremelimumab

INTERVENTIONS:
Drug: CP-675,206 — This is a single arm study. Patients will receive intravenous administration of CP-675,206 at a dose of 15 mg/kg on Day 1 of every 90-day cycle for up to 4 cycles. For purposes of treatment visits and scheduling, each cycle is defined as a 90 (± 4 day) period. Patients who discontinue treatment after 4 doses of CP-675,206 without disease progression and who subsequently experience disease progression more than 3 months after the last dose may receive 2 additional doses of CP-675,206 provided that they have not received other systemic therapy for their melanoma
  Survival in this study will be monitored on all patients for up to 5 years from the date of first dose of CP-675,206.

SUMMARY:
The purpose of this study is to provide access to CP-675,206 for patients with advanced unresectable melanoma and who have the potential to gain benefit from this treatment and who are not eligible for participation in other CP-675,206 studies.

DETAILED DESCRIPTION:
This is an expanded access trial that canceled prior to enrolling patients.

ELIGIBILITY:
Inclusion Criteria:

* Advanced melanoma with life expectancy of at least 6 months.
* Melanoma must be considered unresectable.
* Patients with stable, treated brain mets must be stable clinically and radiographically and off steroids for at least one month.

Exclusion Criteria:

* Patients must not be eligible for participation in any ongoing CP-675,206 clinical studies currently open for enrollment.
* History of chronic inflammatory or autoimmune disease.
* History of inflammatory bowel disease, celiac disease, or other chronic gastrointestinal conditions associated with diarrhea, active colitis, history of diverticulitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-05

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3671028&StudyName=Treatment%20Use%20Study%20for%20Advanced%20Melanoma.